CLINICAL TRIAL: NCT02267252
Title: Effects of Male-specific Antibodies on Sex Ratio
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Consultant, Ph.D., Odense University Hospital
Other Study IDs: Lab.Reprod.Biol.- Odense.01
Record Dates: First submitted 2014-10-08; First posted 2014-10-17 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Sperm Antibodies; Sex Ratio

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and ejaculates
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Antibody-sperm binding

SUMMARY:
Investigation of the ability of antibodies from vasectomized men in binding to Y-spermatozoa as a possible explanation of the lower sex ratio observed after microinsemination using epididymal sperm from vasectomized men.

ELIGIBILITY:
Inclusion Criteria:

* Vasectomized men

Exclusion Criteria:

* Men who do not understand the study information

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Vasectomized men
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Y/X sperm ratio after exposure to sperm-specific antibodies | Up to 28 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fertility Clinic, Odense University Hospital, Odense, Denmark